CLINICAL TRIAL: NCT01317537
Title: Using an Electronic Personal Health Record to Empower Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Cerner Corporation (Unknown); The Institute for Patient- and Family-Centered Care (Other)
Responsible Party: Peggy J Wagner, Georgia Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: HS017234
Record Dates: First submitted 2011-03-02; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: personal health records
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Received personal health record (Experimental): received personal health record access
  Interventions: Other: Electronic personal health record
- No personal health record (No Intervention): did not receive personal health record

INTERVENTIONS:
Other: Electronic personal health record
  Arms: Received personal health record

SUMMARY:
Project Summary:

An electronic personal health record (ePHR) could maximize patient/clinician collaboration and consequently improve patient self-management and related health outcomes. The purpose of the proposed project is to examine the feasibility, acceptability, and impact of an ePHR that has been modified using a patient- and family-centered approach and incorporates the experiences, perspectives, and insights of patients and family members actually using the system. Comparison of patients with the ePHR intervention to a group of "care as usual" patients will be performed. The investigators Specific Aims are: (1) To improve the application of patient- and family-centered care elements in an existing ePHR, based on feedback from a pilot study of patients and their families. The modified ePHR will be tested in a pilot group of patients with hypertension and their families. (2) To implement and test the effectiveness of the modified ePHR with patients being treated for hypertension by a team of physicians, mid-level practitioners, nurse clinicians, and support staff in two ambulatory settings. Outcome measures will include patient activation and perception of care, quantifiable biological markers, patient-physician communication, and congruence of treatment with guidelines, particularly medication management; (3) To monitor the shift in provider and support staff awareness and incorporation of patient- and family-centered care as a result of implementation of the ePHR using questionnaires and focus groups. If successful, this ePHR could be implemented in additional locations in the Southeast.

ELIGIBILITY:
Inclusion Criteria:

* age 21
* hypertension
* referral by physician

Exclusion Criteria:

* age over 80
* no hypertension
* too ill to participate

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 9 months
  2 seated measures taken using manual sphygmometer by trained research associate
Diastolic blood pressure | 9 months
  2 seated measures taken using manual sphygmometer by trained research associate

SECONDARY OUTCOMES:
patient activation | 9 months
  Patients complete the validated paper-and-pencil Patient Activation Measure (PAM) developed by Judy Hibbard. The instrument assesses the degree to which a patient is "activated," that is the degree to which they are an active agent in their own health care, e.g. ask questions of their health care provider.
Patient satisfaction with care | 9 months
  Consumer Assessment of Health care--group and clinician survey Patient assessment of chronic care Post study interviews
adherence to guidelines | 9 months
  chart audit of patient care

CONTACTS AND LOCATIONS:
Overall Officials: Peggy J Wagner, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Wagner PJ, Dias J, Howard S, Kintziger KW, Hudson MF, Seol YH, Sodomka P. Personal health records and hypertension control: a randomized trial. J Am Med Inform Assoc. 2012 Jul-Aug;19(4):626-34. doi: 10.1136/amiajnl-2011-000349. Epub 2012 Jan 10. PMID 22234404